CLINICAL TRIAL: NCT00731055
Title: Effects of Varenicline on Cigarette Self Administration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Adam Bisaga, Research Psychiatrist, New York State Psychiatric Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: #5649/NIDA-17572-4; R01DA017572 (NIH); DPMCDA (Other: NIDA)
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2015-05-01 (Estimated); Last update posted 2018-06-18 (Actual); Status verified 2018-05

CONDITIONS: Nicotine Dependence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Intervention 1 (Experimental): Each participant participates in 4 consecutive interventions in random order.
  1. Placebo, 1 capsule before the session
  2. 0.5 mg varenicline, 1 capsule before the session 3.1 mg varenicline, 1 capsule before the session
  4. 2 mg varenicline, 1 capsule before the session
  Interventions: Drug: Varenicline; Drug: Placebo
- Intervention 2 (Experimental): Each participant participates in 4 consecutive interventions in random order. 1.0.5 mg varenicline, 1 capsule before the session 2. 1 mg varenicline, 1 capsule before the session 3.2 mg varenicline, 1 capsule before the session 4. Placebo, 1 capsule before the session
  Interventions: Drug: Varenicline; Drug: Placebo
- Intervention 3 (Experimental): Each participant participates in 4 consecutive interventions in random order. 1.1 mg varenicline, 1 capsule before the session 2. 2 mg varenicline, 1 capsule before the session 3.Placebo, 1 capsule before the session 4. 0.5 mg varenicline, 1 capsule before the session
  Interventions: Drug: Varenicline; Drug: Placebo
- Intervention 4 (Experimental): Each participant participates in 4 consecutive interventions in random order. 1.2 mg varenicline, 1 capsule before the session 2. Placebo, 1 capsule before the session 3. 0.5 mg varenicline, 1 capsule before the session 4. 1 mg varenicline, 1 capsule before the session
  Interventions: Drug: Varenicline; Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — 4 doses of Varenicline. 1 capsule of either dose (0mg, 0.5mg, 1mg, 2 mg) in the morning on days at least 5 days apart.
  Other Names: Chantix
Drug: Placebo — 1 dose of placebo

SUMMARY:
The investigators hypothesize that varenicline will dose dependently attenuate the subjective effects of cigarettes after a period of abstinence. Also, treatment with varenicline will dose dependently weaken the severity of nicotine withdrawal symptoms. Thirdly, we hypothesize that treatment with varenicline will dose dependently decrease cigarette self-administration in the model proposed.

DETAILED DESCRIPTION:
Tobacco use is the leading preventable cause of death in the U.S.A. Every year 400,000 people die from cigarette smoking and in 2006, one out of every five deaths in the US were smoking related. Recent advances in laboratory studies of tobacco effects in humans and in understanding the effects of nicotine on the brain and behavior present an opportunity to advance medication development.

The addictive properties of nicotine are thought to be a result of nicotine triggering the acute release of dopamine, a pleasurable event that a person seeks to repeat. Varenicline is a partial agonist of the nicotine receptors, therefore also triggering the release of dopamine but in a more sustained and moderate manner, which could counter the low dopamine levels arising from a lack of nicotine and therefore aid craving. Also, by binding to these nicotine receptors in advance of smoking, it could stop nicotine from binding and creating pleasurable effects.

This study will assess the effect of acute treatment with varenicline and placebo on early tobacco withdrawal, acute effects of cigarettes and cigarette self-administration in cigarette-smoking volunteers. After overnight abstinence, participants will come into the lab and receive acute treatment with varying doses of varenicline or placebo and perform computer tests and fill out questionnaires. Then they will be given the opportunity to smoke under operational conditions (cigarette versus money choice). This study will employ a within-group, double-blind, randomized and counterbalanced design.

The main goal of this project is to improve the current laboratory model of smoking cessation and study the mechanism involved in smoking maintenance. We hypothesize that varenicline will dose-dependently: 1) decrease nicotine withdrawal symptoms, 2) decrease acute effects of cigarettes and 3) decrease self-administration of cigarettes in the laboratory paradigm. Showing the effectiveness of varenicline in the proposed laboratory model will confirm the model's predictive validity to detect clinically effective medication.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of nicotine dependence with physiological dependence, smoking at least 15 cigarettes/day during the last 3 months.
2. Not interested in treatment
3. Medically healthy on the basis of physical examination and medical history, vital signs, EKG and laboratory tests, with a negative pregnancy test for females.
4. Able to perform study procedures
5. Males or females between the ages of 21-45 yrs
6. Female participants agree to use an effective method of birth control during the course of the study

Exclusion Criteria:

1. A diagnosis of abuse or dependence on alcohol or drugs other than nicotine
2. Current Axis I diagnosis or current treatment with psychotropic medications (within last 3 months)
3. Lifetime history of schizophrenia or other psychotic disorders, bipolar disorder, or anxiety disorders
4. Currently seeking treatment for nicotine dependence
5. Participants on parole or probation
6. History of significant recent violent behavior
7. Blood pressure > 150/90
8. History of allergic reaction to any of the study medications

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2008-02; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam Bisaga, MD, Principal Investigator — New York State Psychiatric Institute
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Twenty-one participants were recruited in an urban hospital setting through advertisement in local newspapers and flyers and 16 particiopants were enrolled. Study was conducted at the NYS Psychiatric Institute
Groups:
- Study Participants: This is a within-group study design, all participant who completed the study receive all 4 experimental treatments
Period: Overall Study
Arm/Group | Study Participants
Started | 16 (This is a within-subjects study design.)
Received Placebo | 16
Received Varenicline 0.5 mg | 16
Received Varenicline 1.0 mg | 16
Received Varenicline 2.0 mg | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Study Participants: Each of study participants received one dose of study medication (varenicline 0mg, 0.5mg, 1mg, and 2 mg) before each of the experimental sessions at least 5 days apart.
Arm/Group | Study Participants
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 36.5 [23 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 10
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Cigarette Choice
Description: Over each of the four 6-hour experimental sessions, a participant was asked 9 times if they would take money or a cigarette. This outcome measure assesses the number of times a participant chose a cigarette.
Time Frame: During each of the four weekly 6-hour experimental sessions
Measure: Mean (Standard Deviation); unit: number of cigarette choices (0-9)
Groups:
- Placebo: The outcome of the session during which participant received placebo
- Varenicline 0.5 mg: The outcome of the session during which participant received varenicline 0.5 mg
- Varenicline 1.0 mg: The outcome of the session during which participant received varenicline 1.0 mg
- Varenicline 2.0 mg: The outcome of the session during which participant received varenicline 2.0 mg
Arm/Group | Placebo | Varenicline 0.5 mg | Varenicline 1.0 mg | Varenicline 2.0 mg
Number analyzed (Participants) | 16 | 16 | 16 | 16
number of cigarette choices (0-9) | 3.67 (0.51) | 3.17 (0.63) | 2.83 (0.71) | 2.83 (0.55)

ADVERSE EVENTS:
Time Frame: Adverse events reported during 4 experimental sessions
Arm/Group | Study Participants
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes